CLINICAL TRIAL: NCT05634798
Title: An Observational Study Based on Endometrial Cancer Risk Screening Model
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-3525
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-05

CONDITIONS: Endometrial Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — There is no intervention in this study.

SUMMARY:
The goal of this observational study is to test the efficiency of our endometrial cancer risk screening calculator, and improve the endometrial cancer risk screening model to form a stable and reliable non-invasive auxiliary diagnostic tool with high sensitivity and specificity in healthy women.The main question it aims to answer is:

·the efficiency of our endometrial cancer risk screening calculator Participants will be collected demographic information, as well as ultrasound, blood routine test and other test results, which will be entered into the endometrial cancer risk screening calculator to obtain high-risk or low-risk prediction results.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70;
2. The annual update of questionnaire information required by the calculator can be completed, and the gynecological examination, gynecological B-ultrasound and blood test can be evaluated once a year, and the follow-up can be at least 1 year; The patient or family members can understand the research scheme and are willing to participate in the study, and provide e-book informed consent.

Exclusion Criteria:

1. Endometrial cancer or precancerous lesions have been diagnosed;
2. Previous or current malignant tumor, currently receiving radiotherapy and chemotherapy, endocrine, targeted and immunotherapy;
3. History of endometrial resection or total hysterectomy;
4. Pregnant or lactating women;
5. The patient or family member could not understand the conditions and objectives of this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects were women of childbearing age, perimenopause and postmenopausal who had undergone physical examination in Peking Union Medical College Hospital or were recruited by patients from gynecological clinics.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Obtained endometrial pathological specimens due to any factors | 1 year
  The study object was obtained endometrial pathological specimen within one year due to any factor.
No endometrial cancer or precancerous lesions | 1 year
  The study object did not show B-ultrasound and clinical symptoms which indicate endometrial cancer or precancerous lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Shu Wang, Doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No